CLINICAL TRIAL: NCT02960932
Title: Reproducibility Inter-session of the Measurement Elastography of the Passive Stiffness of Medial Beams of Gastrocnemius Muscle of the Hemiplegic Cerebral Child.
Acronym: ELASTOREPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1608112; 2016-A01558-43 (Other: ANSM)
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-03

CONDITIONS: Gait; Child Development; Hemiplegic
Keywords: Hemiplegic; Child; Elastography; paralysis
MeSH Terms: conditions — Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hemiplegic cerebral child (Experimental): Ultrasound scanner used to the SSI technical reproducibility.
  Interventions: Device: ultrasound scanner

INTERVENTIONS:
Device: ultrasound scanner — Ultrasound scanner used to the SSI technical reproducibility.

SUMMARY:
Muscles, paretics and spastics, of cerebral palsy children have very early, for growth (three at five aged), every alteration of theirs properties. Gastrocnemius muscle, often reaches on the cerebral palsy, characterised by a modification of the structure (volume decrease) and the elasticity (increase of the passive stiffness). Every alterations of the muscular property have impact clinic and functional important. The many treatments of orthopaedic targeting (lengthening of cast, injections of botulinic toxin), repeated to a multiple recovery during the growth influences the muscular characteristics. There is a real interest to measure the muscular property development during children's growth.

DETAILED DESCRIPTION:
Elastography is a technical assessment of characteristic of the soft tissues. In this area, the method " Supersonic Shear Imaging® (SSI) " provide an important technological change measuring, swiftly and no invasive, a elasticity modulus reflecting the property visco-elastic of the muscle. A lot of ex vivo study led in isolated muscle and in vivo in healthy adults demonstrated the validity of the method SSI on the evaluation of the passive stiffness from a number of muscle group whose the gastrocnemius muscle. The main objective of this study must be checked the intersession reproducibility of the method SSI on the evaluation of the passive stiffness at the medial bundle of the gastrocnemius muscle therefore their passive lengthening in cerebral palsy children. The secondary objective is to test the correlation level of the relation elasticity modulus/ joint angle and couple force-angle obtained throughout the passive lengthening at the medial bundle of the gastrocnemius muscle in cerebral palsy children.

ELIGIBILITY:
Inclusion Criteria:

* Parents affiliated or entitled to a social security;
* Children diagnosed spastic cerebral paralyzed, with a clinical picture of hemiplegia infantile cerebral;
* Children walking GMFCS (Gross Motor Functional Classification System) between I and III;
* Children with spasticity level in the paralysing gastrocnemius muscle greater than or equal X1, VII, on the scale of Tardieu and 2 on the Ashworth scale.
* Children aged 5 to 12 years.
* Children can understand and follow the simple instructions in the examination process.
* Consent signed by the holder of parental authority.

Exclusion Criteria:

* Children with concomitant muscle disease (myopathy ...).
* Children who received another treatment to target relaxant (baclofen, ... muscle relaxant) which would have begun in the months preceding the assessment.
* Children who underwent neuro-orthopedic surgery at the where paretic members.
* Children who received an injection of botulinic toxin for less than 15 days.
* Children who have benefited from extensions casts for less than 7 days.
* Children who received a therapeutic target for orthopedic (botulinum toxin, plaster of extensions, installation of equipment of lower limb) between the two sessions evaluations.
* Children who received a physiotherapy session the day before evaluation elastography and ultrasound.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Measure of elasticity modulus | 7 days
  To measure at the medial bundle of the gastrocnemius muscle at the passive mobilization of the ankle in the joint sector following: 30 degree in plantar and maximal dorsal flexion; calculation of yield curve of elasticity modulus, joint angle in kilopascals (kPa).

SECONDARY OUTCOMES:
Measure of force couple | 7 days
  Stored measure at the passive mobilization of the ankle in position of maximal dorsal flexion; calculation of yield couple of joint force-angle in nanometer.
Measure of fascicular length | 7 days
  To measure at the medial bundle of the gastrocnemius muscle at the passive mobilization of the ankle in the selected joint sector (30 degree in plantar and maximal dorsal flexion); calculation of the difference of fascicular length in millimeter between the extreme position of joint sector: 30 degree in plantar and maximal dorsal flexion.
Measure of pennation angle of the muscular fascicle | 7 days
  To measure at the medial bundle of the gastrocnemius muscle at the passive mobilization in the selected joint sector in degree; calculation of the difference of pennation angle of the muscular fascicle between the extreme position of joint sector: 30 degree in plantar and maximal dorsal flexion.
Measure of elasticity modulus | 7 days
  Measure of elasticity modulus at the medial bundle of the gastrocnemius muscle in rest position kilopascals (kPa).
Measure of muscle stiffness | 7 days
  Difference of muscle stiffness evaluated between the paretic and no paretic member.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gautheron, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boulard C, Gautheron V, Lapole T. Reliability outcomes and inter-limb differences in ankle joint stiffness in children with unilateral cerebral palsy depend on the method of analysis. J Electromyogr Kinesiol. 2019 Dec;49:102353. doi: 10.1016/j.jelekin.2019.102353. Epub 2019 Aug 23. PMID 31473451